CLINICAL TRIAL: NCT07376408
Title: The Effect of Spousal Support on Sexual Quality of Life in Postmenopausal Women
Brief Title: Spousal Support and Sexual Quality of Life in Postmenopausal Women
Status: Not yet recruiting | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Eslem Altıntaş, MSc, Acibadem University
Other Study IDs: 2026/02
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Postmenopausal; Support; Sexuality
Keywords: Postmenopausal; Sexuality; Quality of Life; Support
MeSH Terms: conditions — Sexuality

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Postmenopausal Women: Postmenopausal women with a partner, registered at Family Health Centers in Istanbul, who participate in this observational study to assess perceived spousal support and sexual quality of life. No intervention is applied.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is an observational study. No intervention, treatment, or behavioral modification is applied. Data are collected using self-reported questionnaires only.

SUMMARY:
Menopause is a natural transition period in women's lives characterized by concurrent hormonal, psychological, and relational changes. During the postmenopausal period, hormonal alterations are not limited to physical symptoms but also have significant effects on psychological well-being, interpersonal relationships, and particularly sexual quality of life. Common concerns during this period include decreased sexual desire, vaginal dryness, pelvic discomfort, and reduced sexual satisfaction, all of which may negatively affect overall quality of life. Sexual quality of life is influenced not only by biological factors but also by psychological and relational dimensions.

The quality of partner relationships and perceived partner support play an important role in women's adaptation to sexual changes during the postmenopausal period. However, partner support during menopause is often reported to be insufficient, which may adversely affect sexual well-being. Despite this, evidence examining the relationship between perceived partner support and sexual quality of life in postmenopausal women remains limited.

The aim of this study is to examine the effect of perceived partner support on sexual quality of life in postmenopausal women. Through this investigation, the explanatory role of partner support in postmenopausal sexual well-being is aimed.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal status, defined as at least 12 consecutive months of amenorrhea
* Having a partner
* Voluntary agreement to participate in the study and provision of written informed consent

Exclusion Criteria:

* Visual, cognitive, or other impairments that prevent completion of the study questionnaires
* History of major gynecological surgery within the past 6 months

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population consists of postmenopausal women registered at Family Health Centers in Istanbul, Türkiye. Eligible participants are women who are in the postmenopausal period, defined as having experienced at least 12 consecutive months of amenorrhea, who have a partner, and who voluntarily agree to participate in the study. Data will be collected using self-reported questionnaires, and no intervention will be applied.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Introduction Information Forum | At enrollment
  This form was developed by the researchers based on the relevant literature and consists of 36 items assessing participants' sociodemographic and clinical characteristics, including age, educational level, employment status, duration of marriage, duration of menopause, and presence of chronic disease.
The Sexual Quality of Life-Female Questionnaire | At enrollment
  The Sexual Quality of Life-Female Questionnaire (SQoL-F) was developed by Symonds et al. (2005) to assess women's perceived sexual quality of life. The Turkish validity and reliability study was conducted by Tugut and Golbasi (2010).
  The scale consists of 18 items, each rated on a 6-point Likert scale (1 = Completely agree, 6 = Completely disagree). The raw total score ranges from 18 to 108. Items 1, 5, 9, 13, and 18 are reverse scored prior to calculating the total score.
  The raw total score is transformed to a 0-100 scale using the following formula:
  (raw score - 18) × 100 / 90.
  Higher scores indicate better sexual quality of life, whereas lower scores indicate poorer sexual quality of life. The Cronbach's alpha coefficient of the Turkish version is reported as 0.83.
The Menopause Spousal Support Scale | At enrollment
  The Menopause Spousal Support Scale was developed to assess perceived spousal support among women during menopause. The Turkish validity and reliability study was conducted by Küçükkelepçe et al. (2024).
  The scale consists of 17 items and includes four subscales: emotional support, instrumental support, esteem support, and sexual intimacy support. Items are rated on a 10-point Likert scale ranging from 1 (never) to 10 (almost always).
  The total score ranges from 17 to 170. Higher scores indicate greater perceived spousal support, whereas lower scores indicate lower perceived spousal support. The Cronbach's alpha coefficient of the Turkish version is 0.96.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Coşkun, Ph.D., Principal Investigator — Acibadem University; Nevin Şahin, Prof. Dr., Principal Investigator — Istanbul University-Cerrahpaşa, Institute of Graduate Studies, PhD Program
Locations (1):
- Istanbul Provincial Directorate of Health - Family Health Centers, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No